CLINICAL TRIAL: NCT06597461
Title: Acute Effects of Myofascial Release on Foot Mobility and Performance in Basketball Players With Hypomobile feet-a Randomized Controlled Trial
Brief Title: Myofascial Release and Foot Mobility in Basketball Players: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, Nihat Sarıalioğlu, Assistant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRU-SBF-NS-01
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Foot Deformities
Keywords: hypomobile feet; basketball players; myofascial release; foot mobility; performance
MeSH Terms: conditions — Foot Deformities | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: Two groups with a control group
Who Masked: Participant
Masking Description: Participants were not informed which group they were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial release (MR) group (Active Comparator): The group that received Graston myofascial application
  Interventions: Other: Myofascial release
- Placebo myofascial release (PMR) group (Placebo Comparator): The group that received placebo Graston myofascial application
  Interventions: Other: Placebo myofascial release

INTERVENTIONS:
Other: Myofascial release — Graston massage technique was used in the application. In the application, the participant was placed in a prone position and the feet were left slightly outside the massage table. The application was performed on the entire plantar surface between the calcaneal tuberosity and metatarsophalangeal joints in the form of multidirectional strokes at 30-60 degrees with the GT 4 graston tool. The total application took an average of 5 minutes for each foot. An average of 60-70 strokes were performed per minute and 10 seconds of rest was given every minute. The application was performed as a single session by an expert physiotherapist.
  Other Names: Placebo myofascial release
  Arms: Myofascial release (MR) group
Other: Placebo myofascial release — Graston massage technique was used in the application. In the application, the participant was placed in a prone position and the feet were left slightly outside the massage table. The application was performed on the entire plantar surface between the calcaneal tuberosity and metatarsophalangeal joints in the form of multidirectional strokes at 30-60 degrees with the GT 4 graston tool. The total application took an average of 5 minutes for each foot. An average of 60-70 strokes were performed per minute and 10 seconds of rest was given every minute. The application was performed as a single session by an expert physiotherapist. Since it was a placebo application, no pressure was applied to the tissues by the physiotherapist during the strokes.
  Arms: Placebo myofascial release (PMR) group

SUMMARY:
The purpose of this study was to investigate the acute effects of myofascial release on foot mobility and sportive performance in basketball players with hypomobile feet. This study was designed as randomized controlled experimental research.

DETAILED DESCRIPTION:
Hypomobility in the foot structure causes functional limitations. These functional limitations affect the sportive performance negatively, especially in basketball where dynamic movements such as jumping and sudden change of direction are very intense. In this context, reducing hypomobility is important in terms of eliminating performance disorders caused by hypomobility. The purpose of this study was to investigate the acute effects of myofascial release on foot mobility and sportive performance in basketball players with hypomobile feet. This study was designed as randomized controlled experimental research. Twenty-four male basketball players (23.46±2.81 years) participated in the study. Athletes were first subjected to foot mobility, balance and vertical jump tests. Then the participants were divided into two groups as myofascial release (MR) and placebo myofascial release (PMR). Myofascial release was applied to the MR group and placebo myofascial release was applied to the PMR group. After the application, foot mobility and performance measurements were performed again and the results were analyzed. It was observed that there was a significant difference in right foot mobility (RFM), left foot mobility (LFM), vertical jump (VJ) and dynamic balance (DB) parameters after the application in MR group (p<0.001), while there was no change in any parameter after the application in PMR group (p>0.05). The results of this study show that a single session of myofascial release applied to the plantar sole temporarily increased foot mobility and improved vertical jump and dynamic balance performance in basketball players with chronic hypomobility.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players who had hypomobility in at least one foot, had not had a serious foot or ankle injury in the last year, and had been actively licensed for the last five years were included in the study.

Exclusion Criteria:

* Those who did not meet the inclusion criteria were excluded from the study.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-17 (Actual)

PRIMARY OUTCOMES:
hypomobility measurement | 6 hours
  Therefore, firstly, the degree of foot mobility of all participants was measured, and height and body weight measurements the balance characteristics and vertical jump levels of the participants who met the inclusion criteria were determined. TParticipants were not informed which group they were in. The MR group received myofascial release and the PMR group received placebo (superficial) myofascial release. All myofascial release applications were performed by an expert physiotherapist. After the application, the degree of foot mobility, balance characteristics and vertical jump levels of the participants were measured again. In order to determine the duration of the acute effects of mobility after myofascial release, the MR group was subjected to a 2-hour standard basketball training after the second measurements. Foot mobility was measured three more times at one-hour intervals in the first hour of the training, at the end of the training and then at rest.

SECONDARY OUTCOMES:
Height and body weight measurements | 4 hours
  The height measurements of the participants were measured with wall-mounted holtain stadiometer and body weight and body mass index (BMI) measurements were measured with Tanita MC-580 body analyzer.
Evaluation of foot mobility | 4 hours
  The modified navicular drop (MND) test was used to assess foot mobility. The MND test is an easy, valid and clinical method used in the evaluation of foot mobility. In the navicular drop test, the navicular process was palpated externally while the subject was sitting on a chair with the foot in neutral position and the height above the ground was measured. The subject was then made to stand up and place one foot on a specially designed 10.16 cm (4 inch) high box without weight. The height above the ground of the navicular process of the loaded foot was measured again. Feet with a difference of less than 4 mm between unweighted and weighted measurements were recorded as hypomobile. The reference values of navicular mobility in the MND test are 0-4 mm hypomobile foot, 5-9 mm neutral foot and 10 mm or more hypermobile foot.
Vertical jump measurements | 4 hours
  Vertical jump values were performed with arm swing countermovement jump technique using smart speed brand electronic jump mat. The athlete took a position on the jumping mat with feet one shoulder length apart. Then, when he felt ready, he stretched downward and jumped vertically to the highest point he could jump and fell back on the mat. Three attempts were made in the correct position, 3 seconds rest time was allowed between each jump, and the best degree was recorded in cm. The jumps were repeated with the knees flexed while the athlete remained in the air.
Determination of balance levels | 4 hours
  The balance score was calculated by summing the standard deviation of the front-to-back swing and the standard deviation of the right-to-left swing. The multiaxial proprioceptive assessment module of the isokinetic measurement system was used to determine the dynamic balance levels. First, the device was calibrated and the system was introduced to the volunteers. The volunteers' feet were placed on the platform with reference to the x and y lines on the platform. In the measuring position, the hands were drooping and the feet were bare. Measurements were made in bipedal and 10 difficulty levels for 60 seconds. The test was stopped and restarted when situations such as falling or touching any part of the device occurred during the measurement. Dynamic balance levels were assessed using the average tracking error (ATE).
Myofascial release application | 4 hour
  Graston massage technique was used in the application. In the application, the participant was placed in a prone position and the feet were left slightly outside the massage table. The application was performed on the entire plantar surface between the calcaneal tuberosity and metatarsophalangeal joints in the form of multidirectional strokes at 30-60 degrees with the GT 4 graston tool. The total application took an average of 5 minutes for each foot. An average of 60-70 strokes were performed per minute and 10 seconds of rest was given every minute. The application was performed as a single session by an expert physiotherapist.

CONTACTS AND LOCATIONS:
Overall Officials: Nihat SARIALİOĞLU, PhD, Principal Investigator — Giresun University
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No